CLINICAL TRIAL: NCT05204667
Title: Efficacy and Safety of Different Dosage Regimens of the Combination Methocarbamol/Paracetamol in Acute Low Back Pain (LBP): MioPain Study
Brief Title: Different Dosage Regimens of Methocarbamol/Paracetamol in Acute Non-specific Low Back Pain. MioPain Study
Acronym: MioPain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study had to be closed because it was not feasible to reach the estimated sample size.
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 044(10A)MD20294; 2021-000067-68 (EudraCT Number)
Record Dates: First submitted 2021-12-14; First posted 2022-01-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: low back pain; methocarbamol; paracetamol; Robaxisal compuesto
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a Phase IV, randomized, open-label, parallel-group, multicentre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methocarbamol 380 mg/paracetamol 300 mg (4 times/day) (Experimental): Patients treated with two oral tablets of methocarbamol 380 mg/paracetamol 300 mg 4 times/day up to 7 days (i.e., every 6 hours±1 hour).
  Interventions: Drug: 380 mg/300 mg comprimidos metocarbamol/paracetamol - 4 times daily
- Methocarbamol 380 mg/paracetamol 300 mg (6 times/day) (Active Comparator): Patients treated with two oral tablets of methocarbamol 380 mg/paracetamol 300 mg 6 times/day up to 7 days (i.e., every 4 hours±1 hour).
  Interventions: Drug: 380 mg/300 mg comprimidos metocarbamol/paracetamol - 6 times daily

INTERVENTIONS:
Drug: 380 mg/300 mg comprimidos metocarbamol/paracetamol - 4 times daily — (2 oral tablets 4 times/day up to 7 days (i.e., every 6 hours±1 hour). Ingestion of the tablets can be helped with a small amount of water.
  Other Names: Robaxisal compuesto
  Arms: Methocarbamol 380 mg/paracetamol 300 mg (4 times/day)
Drug: 380 mg/300 mg comprimidos metocarbamol/paracetamol - 6 times daily — (2 oral tablets 6 times/day up to 7 days (i.e., every 4 hours±1 hour). Ingestion of the tablets can be helped with a small amount of water.
  Other Names: Robaxisal compuesto
  Arms: Methocarbamol 380 mg/paracetamol 300 mg (6 times/day)

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of different dosage regimens of the combination methocarbamol/paracetamol in the treatment of patients with acute non-specific Low Back Pain.

DETAILED DESCRIPTION:
This is a Phase IV, randomized, open-label, parallel-group, multicentre study.

A total of 192 patients of both sexes will be enrolled in the study and will be randomized 1:1 to one of the following 2 treatment groups:

* Group 1: methocarbamol 380 mg/paracetamol 300 mg (2 oral tablets 4 times/day)
* Group 2: methocarbamol 380 mg/paracetamol 300 mg (2 oral tablets 6 times/day) The expected duration of patient participation into the trial (from ICF signature up to any applicable follow up) is 8 days (± 1). Patients enrolment will be competitive among clinical sites.

The primary endpoint will be the Time to complete relief of pain, defined as the time when the complete pain relief is reached. A Complete pain relief is defined as a VAS score ≤ 5 mm at two consecutive assessments starting from Day1 up to Day7 (±1).

ELIGIBILITY:
Inclusion Criteria:

-Male and female patients of any ethnic origin between 18 and 64 years of age (limits included).

-Patients with current episode of acute (pain lasting less than 6 weeks) non-specific LBP, defined as pain and discomfort, localised below the costal margin and above the inferior gluteal folds, with or without leg pain, or acute exacerbation of chronic low back pain defined with a VAS score ≥ 40 mm.

* Patients with signs and symptoms of muscle spasm of the lumbar region, as clinically diagnosed by the Investigator.
* Women of childbearing potential and women with no menses for a period < 12 months must have a negative pregnancy test at Visit 0 and have to agree not to start a pregnancy from the signature of the informed consent up to the Final Visit/Visit 2, using an appropriate birth control method such as combined oestrogen-progestin containing hormonal contraceptives (e.g., oral, injectable, transdermal), progestin-only hormonal contraceptives (e.g., oral, injectable, implantable), intrauterine device (IUD) or Intrauterine hormone-releasing System (IUS) in combination with male condom, bilateral tubal occlusion, vasectomised partner, sexual abstinence. The following definitions will be considered:
* Woman of childbearing potential (WOCBP): i.e., fertile, following menarche and until becoming post-menopausal, unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.
* A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Patients legally capable of giving their consent to participate in the study and available to sign and date the written Informed Consent.

Exclusion Criteria:

-1. Known hypersensitivity or allergy to the active ingredients and/or to any component of the study medications.

2. Lactating and pregnant women. 3. Clinically significant abnormalities on physical examination and vital signs at Visit 0 which in the opinion of the Investigator could interfere with the study procedures or endpoints evaluation.

4. Suspicious (according to the patient's symptoms at baseline) or confirmed COVID-19 infection at time of screening visit.

5. History of cervical, thoracic, or lumbosacral pain for ≥75% of the time in the last year, or any other LBP episode in the last 3 months that required pharmacological treatment with an opioid analgesic.

6. Patients with:

* serious spinal pathology; spinal surgery in the year prior to screening or history of more than one spinal surgery; history of severe lumbar spinal stenosis; ankylosing spondylitis; lumbosciatalgia; herniated disc or radiculopathy; severe arthritis and osteoporosis; muscular diseases, such as myositis, poliomyelitis, muscular dystrophy and myotonia; fibromyalgia; myasthenia grave; fracture or recent history of violent trauma of the back; structural deformity of the back;
* cancer, not in remission or in complete remission less than 1 year;
* active influenza or other viral syndrome; immunosuppression; systematically unwell; unexplained significant weight loss;
* women with polymenorrhea, endometriosis, ovarian cysts, uterine fibroids;
* widespread neurological symptoms (including cauda equina syndrome) or any brain disease; ever suffered from any brain damage or have been in a coma; epilepsy or seizures;
* active or suspected esophageal, gastric, pyloric channel, or duodenal ulceration, or bleeding in the last 30 days;
* previous treatment with anticoagulants in the seven days before the screening visit;
* renal and/or hepatic failure;
* acute hepatitis;
* cardiac or pulmonary diseases;
* acetylsalicylic acid-triggered asthma;
* glucose-6-phosphate dehydrogenase-deficient patients; glutathione deficiency, dehydration, chronic malnutrition; anemia.

Any other condition that, in the opinion of the Investigator, interferes with the study endpoints/procedures and does not justify the inclusion of the patient in the study.

7. Current use of full, regular, recommended doses of any skeletal muscle relaxants/non - opioid analgesics/anti-inflammatory/NSAIDs in the 6 hours prior to the screening visit. Use is forbidden for the entire trial duration.

8. Current use of full, regular, recommended doses of or any medication that can alter the perception of pain (e.g., opioids, heparinoids, psychotropic agents, anti-H1 agents or glucocorticosteroids, etc.), in the 24 hours prior to the screening visit. Use is forbidden for the entire trial duration.

Chronic intake of low doses of acetylsalicylic acid, i.e., ≤162 mg/daily, taken for at least 30 days prior to the first dose of study medication for non-analgesic reasons could be continued for the duration of the study.

9. Current use of the following medications (use is forbidden for the entire trial duration):

• systemic corticosteroids;

* other drugs containing paracetamol;
* central nervous system (CNS) depressants and stimulants, including barbiturates, anaesthetics, appetite suppressants, anticonvulsants and lamotrigine (with the exception of therapeutic doses of benzodiazepines used as hypnoinducers in patients stabilised for more than one month since the screening visit);
* anticholinergic drugs; psychotropic drugs; anti-cholinesterase drugs, pyridostigmine;
* oral anticoagulants;
* chloramphenicol; rifampicin; zidovudine;
* loop diuretics;
* isoniazid; probenecid;
* propranolol;
* antiemetics;
* metoclopramide; domperidone;
* ion exchange resins (e.g. cholestyramine).

  10. Patients undergoing physiotherapy, osteopathy or chiropractic treatments aimed to reduce LBP.

  11. Patients treated with invasive procedures aimed to reduce LBP (e.g., epidural injections, spinal cord stimulation therapy).

  12. History of alcoholic/substance abuse. Use of alcohol is forbidden during the entire duration of the study.

  13. Inability to comply with the protocol requirements, instructions or study-related restrictions (i.e., uncooperative attitude, inability to return for study visits, unlikelihood of completing the clinical study); vulnerable patients (i.e., persons kept in detention).

  14. Patients involved in the conduct of the study (i.e., Investigator or his/her deputy, first grade relatives, pharmacist, assistant or other personnel).

  15. Participation to an interventional clinical trial within 3 months prior to Visit 0.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Time to complete releif of pain. | from Day1 up to Day7 (±1).
  The Time to complete relief of pain is defined as the time when the complete pain relief is reached.
  A Complete pain relief is defined as a Visual Analogue Scale score ≤ 5 mm at two consecutive assessments starting from Day1 up to Day7 (±1).

SECONDARY OUTCOMES:
Change in Low Back Pain intensity at Visit 0 and Visit 1 | Day 0 and Day 4 (±1).
  Change in Low Back Pain intensity at Visit 0 and Visit 1, measured by 0-10 cm (100 mm) Visual Analogue Scale, stretching from 0 "no pain" to 10 "pain as bad as it could be".
Change in Low Back Pain intensity at Visit 0 and Final Visit | Day 0 and Day 8 (±1).
  Change in Low Back Pain intensity at Visit 0 and Final Visit, measured by 0-10 cm (100 mm) Visual Analogue Scale, stretching from 0 "no pain" to 10 "pain as bad as it could be".
Change in the degree of improvement in the hand-to-floor distance | Day 0, Day 4 and Day 8 (±1).
  The Hand-to-floor distance, also called fingertip-to-floor test or mobility assessment is the vertical distance between the tip of the middle finger and the floor measured by a simple cm graduated bar (0 value at floor).
  The patient will be asked to bend forward as far as possible and try to touch the floor with his/her fingers, while maintaining the knees, arms, and fingers fully extended.
Change in the functional disability | Day 0, Day 4 and Day 8 (±1).
  The Functional disability is assessed by the Oswestry Disability Index (ODI) that allows to obtain information on how acute Low Back Pain affects ability to manage patients Activities of Daily Living (ADL).
  The Oswestry Disability Index contains 10 sections. For each section the total possible score is 5: if the first statement is marked, the section score is=0; if the last statement is marked, it is=5. The total score of all sections as a percentage of the total achievable score is the Oswestry Disability Index score.
Change in the Patients' Global Impression of Change scale score | Day 0 and Day 8 (±1).
  The Patients' Global Impression of Change (PGIC) scale reflects a patient's belief about the efficacy of treatment evaluating all aspects of patient's health and quality of life (QoL).
  It is a 7-point scale depicting a patient's rating of overall improvement: "no change", "almost the same", "a little better", "somewhat better", "moderately better", "better", or "a great deal better".
Change in the Clinical Global Impression-Improvement scale score | Day 0 and Day 8 (±1).
  The Clinical Global Impression-Improvement (CGI-I) scale provides an overall clinician-determined summary evaluation of the treatment.
  It is a 7-point scale: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from the initiation of treatment; 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Monitoring frequency of adverse events (AEs) | 8 (±1) days
  Safety will be assessed by monitoring the frequency of adverse events in each treatment group.
  All AEs will be coded using MedDRA (Medical Dictionary for Regulatory Activities).

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Azienda Sociosanitaria Ligure N. 1, Sanremo, Imperia
  - Azienda Sanitaria Locale Asl Al, Alessandria
  - Azienda Sociosanitaria Ligure Asl 3, Genova